CLINICAL TRIAL: NCT03379649
Title: Platelet Rich Plasma for Patients With Recurrent Implantation Failure: A Prospective Randomized Pilot Study
Brief Title: Platelet Rich Plasma for Patients With Recurrent Implantation Failure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lusine Aghajanova, Assistant Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43265
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Infertility
Keywords: Recurrent implantation failure
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Patients will be blinded to the treatment they received, but providers and investigators will be aware.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PRP (Experimental): Patient with recurrent implantation failure who receives intrauterine infusion of platelet rich plasma
  Interventions: Combination Product: Platelet rich plasma
- Placebo (Placebo Comparator): Patient with recurrent implantation failure who receives intrauterine infusion of embryo culture media
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Platelet rich plasma — Patients will have 60ml of blood drawn. Platelet rich plasma will be obtained by placing the blood in the Arteriocyte Magellan device. 0.5ml of Platelet rich plasma will be placed into the uterus at least 48 hours prior to embryo transfer.
  Arms: PRP
Combination Product: Placebo — Patients will have 60ml of blood drawn. 0.5ml of embryo culture media (the placebo) will be placed into the uterus at least 48 hours prior to embryo transfer.
  Arms: Placebo

SUMMARY:
Patients with recurrent implantation failure are among the most difficult patients to treat, with no proven standard treatment. Platelet rich plasma stimulates cellular processes involved in endometrial regeneration, and in a small case series has shown efficacy for this patient population. We hope to conduct a randomized controlled pilot study to determine whether PRP is indeed an effective treatment for recurrent implantation failure.

DETAILED DESCRIPTION:
Patients considered to have recurrent implantation failure will undergo randomization to receive intrauterine infusions of platelet rich plasma or a placebo of embryo culture media prior to their embryo transfer. All patients will undergo a blood draw to obtain 60ml of blood from which 0.5ml of platelet rich plasma will be obtained. Those randomized to receive the platelet rich plasma will have platelet rich plasma placed into the uterine cavity at least 48 hours prior to the embryo transfer, while those randomized to receive placebo will have embryo culture media placed into the uterine cavity at the same point in time. Those randomized to the placebo group will have the opportunity to be placed into the treatment group if no pregnancy was attained. Transfer outcomes including implantation rate, pregnancy rate, and live birth rate, will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All women who have undergone 3 or more embryo (blastocyst stage) transfers without establishing a clinical pregnancy or 2 or more euploid embryo transfers without establishing a clinical pregnancy, aged 18 - 45, with a normal uterine cavity established within 12 months by hysteroscopy or saline infusion sonogram, planning in vitro fertilization with an embryo transfer at Stanford Fertility and Reproductive Health. The planned transfer must consist of any of the following: a PGS proven euploid embryo, a good quality blastocyst from a patient younger than 37, or a donor oocyte blastocyst.

Exclusion Criteria:

* Abnormal uterine cavity, planning in vitro fertilization with use of a gestational carrier. patients enrolled in other experimental interventions for RIF will be excluded. Patients with only poor quality or cleavage stage embryos.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 10 months following transfer
  Live birth/embryo transfer

SECONDARY OUTCOMES:
Pregnancy | 9 days following transfer
  Positive pregnancy test/embryo transferred

CONTACTS AND LOCATIONS:
Overall Officials: Lusine Aghajanova, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Fertility and Reproductive Health, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nazari L, Salehpour S, Hoseini S, Zadehmodarres S, Ajori L. Effects of autologous platelet-rich plasma on implantation and pregnancy in repeated implantation failure: A pilot study. Int J Reprod Biomed. 2016 Oct;14(10):625-628. PMID 27921085
- [Derived] Aghajanova L, Strug M, Zhang J, Lathi RB. Intrauterine platelet-rich plasma infusion for recurrent implantation failure: a pilot randomized controlled single-blinded clinical trial in the USA. J Assist Reprod Genet. 2025 Nov 17. doi: 10.1007/s10815-025-03752-7. Online ahead of print. PMID 41247443